CLINICAL TRIAL: NCT00230451
Title: A Phase II Trial of Preoperative Chemotherapy and Radiation Therapy Followed by Adjuvant Combination Chemotherapy for Patients With Loco-Regional Esophageal Carcinoma
Brief Title: Pre-operative Chemotherapy and Radiation Therapy for Esophageal Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Susan G. Urba, M.D., University of Michigan
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 9740
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2010-01-15 (Estimated); Status verified 2010-01

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Radiation; Paclitaxel; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Radiation
Drug: Paclitaxel
Drug: Cisplatin
Drug: 5-Fluorouracil

SUMMARY:
Surgery (esophagectomy or removal of the esophagus)has been the standard treatment for cancer of the esophagus. However, evidence suggests that preoperative chemotherapy and radiation therapy may add benefit. The purpose of this study is to determine if a treatment program of combined chemotherapy and radiation therapy prior to surgery and chemotherapy after surgery will delay or eliminate recurrence of the cancer.

ELIGIBILITY:
Patient Eligibility:

1. Histologically confirmed squamous cell carcinoma, adenocarcinoma, or mixed adeno/squamous of the the esophagus or gastroesophageal junction.
2. Disease limited to the esophagus and regional lymph nodes. However, celiac node enlargement will be acceptable for tumors of the distal esophagus, because they will be included in the radiation field.
3. Disease must be able to be encompassed in a single radiation field.
4. No medical contraindication to surgery.
5. All treatment is to be administered at the University of Michigan Medical Center
6. Karnofsky Performance Status > 60%
7. Ages 18-75
8. Adequate renal function (BUN <1.5 x N; creatinine <1,5 mg/dl, or measured creatinine clearance>60 ml/min.).
9. Adequate bone marrow reserve (WBC>3500/ul; Platelets>100,000/ul.).
10. Adequate hepatic function (Bilirubin<1.5x N; AST <2 x upper limit of normal).
11. Prior malignancy is acceptable if the patient is considered to be cured. In most cases this will mean a 5 year disease-free period.
12. Ability to give informed consent.

Exclusion Criteria:

1. Patients with active infection, pregnancy, lactating females, serious inter-current medical conditions including congestive heart failure, cardiac arrhythmias, or symptomatic coronary artery diseases are ineligible.
2. No prior treatment allowed. No prior thoracic radiation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-11; Primary Completion 1999-12 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
To determine the rate of complete histologic response induced by this neoadjuvant chemotherapy and radiation therapy regimen.

SECONDARY OUTCOMES:
To determine the overall survival and time to relapse in patients treated with preoperative chemotherapy and radiation therapy followed by adjuvant combination chemotherapy.
To assess the qualitative and quantitative toxicities of this regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Urba, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States